CLINICAL TRIAL: NCT01454167
Title: Acid Base and Electrolytes Patterns in Drains of Different Operational Wounds and Its Relation to Specific Infections and Seroma Formation
Brief Title: Acid Base and Electrolytes Patterns in Drains Operational Wounds and Its Relation to Complications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Yaron Har-Shai, professor, Carmel Medical Center
Other Study IDs: CMC-13-0130-CTIL
Record Dates: First submitted 2011-10-14; First posted 2011-10-18 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Wounds; Infections; Seroma
Keywords: vacum drains; operational wounds; infections; seroma; acid base; glucose; lactate
MeSH Terms: conditions — Wounds and Injuries; Infections; Seroma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objective- The purpose of this study is to evaluate a connection between PH,PCO2,HCO3,PO2,Na,K,Glu and Lactate patterns in vacuum drains of different plastic operational wounds and its relation to infections and seroma formation.

DETAILED DESCRIPTION:
our objective is evaluation of a connection between PH,PCO2,HCO3,PO2,Na,K,Glu and Lactate patterns in vacum drains of different plastic operational wounds and its relation to infections and seroma formation.

it is possible that early changes in this values might point out an infection or seroma formation of a wound before clinical signs appear.

ELIGIBILITY:
Inclusion Criteria:

* all post operational patients who have a vacum drain/s

Exclusion Criteria:

* patients who are unable to sign a Consent Form (demented,Alzheimer's disease ...)
* patients who refuse participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all post operational patients who have a vacuum drain/s
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Histological confirmation | end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nir Gal Or, Dr, Principal Investigator — carmel medical center- ISRAEL
Locations (1):
- Carmel Medical Center, Haifa, Israel